CLINICAL TRIAL: NCT03813901
Title: Advaita Vedanta and Counselling for Women Who Have Experienced Intimate Partner Violence: Impact on Women's Health
Brief Title: Impact of 'Samalochana' Program on Women Who Have Experienced Intimate Partner Violence (IPV)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NMP Medical Research Institute (Other)
Collaborators: Warwick Research Services (Other); Arsha Vidya Study Centre, Tamilnadu, India (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NMP/Arsha 2091
Record Dates: First submitted 2019-01-21; First posted 2019-01-23 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-01

CONDITIONS: Domestic Violence; Intimate Partner Violence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Samalochana Counselling group (Experimental): Arsha Vidya advaita vedanta based counselling were given to the women
  Interventions: Other: Samalochana Counselling
- Wait-list control group (Other): Wait list group were not given any supportive care during the period. After that, they were offered the similar program as Counselling group.
  Interventions: Other: Wait list control

INTERVENTIONS:
Other: Samalochana Counselling — Counselling program was individual, based on advaita vedanta and traditional philosophical grounds to answer individual fears, concerns,conflicts and difficulties in order to cope and recover.
  Arms: Samalochana Counselling group
Other: Wait list control — Wait list had no intervention offered during the study period. Afterwards, they were offered the counselling for the same duration.
  Arms: Wait-list control group

SUMMARY:
Violence has immediate effects on women's health, which in some cases, is fatal. Physical, mental and behavioural health consequences can also persist long after the violence has stopped. Violence against women and girls occurs in every country and culture and is rooted in social and cultural attitudes and norms that privilege men over women and boys over girls.

Research consistently finds that the more severe the abuse, the greater its impact on women's physical and mental health. In addition, the negative health consequences can persist long after abuse has stopped.Present work shares the impact of arsha vidya counselling for women who has been victim of violence.

ELIGIBILITY:
Inclusion Criteria:

* Woman
* Able to attend regular counselling
* Planning to remain in area for next 6 months
* have experience intimate partner violence (physical, emotional, psychological, and/or sexual), including coercive control from a current or former partner in the previous 12 months and no later than 3 years.

Exclusion Criteria:

* Man
* Under 19 years of age
* Cannot attend at regular basis
* Living outside of the selected study sites, or planning to relocate in next 4 months
* Separated more than 3 years ago

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 102 (Actual)
Dates: Start 2018-06-21 (Actual); Primary Completion 2018-11-22 (Actual); Study Completion 2018-12-21 (Actual)

PRIMARY OUTCOMES:
Change in Quality of Life | Change from baseline to 12-week
  Quality of Life was measured using SF-36 questionnaire

SECONDARY OUTCOMES:
Change in Anxiety | Change from Baseline to 12-weeks
  Anxiety was measured using Beck Anxiety Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Neha Sharma, PhD, Principal Investigator — Warwick Research Services; Buddhatmananda Saraswati, Study Chair — Arsha Vidya Study Centre, India; Vandana Mishra, Study Director — Sarvatra International, South Africa
Locations (1):
- Divya, Jaipur, Rajasthan, India

IPD SHARING:
Plan to Share IPD: Undecided